CLINICAL TRIAL: NCT00386802
Title: ANTIVORIFUNGOL:Strategy of Antifungal Use in Oncohematological Neutropenic Patients. Use of Voriconazole as Early Treatment.
Brief Title: Antifungal Use in Oncohematological Neutropenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004973-55; ANTIVORIFUNGOL
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Invader Fungal Infection
Keywords: Neutropenia; Antifungals
MeSH Terms: conditions — Neutropenia | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Antifungal drug. VORICONAZOL. (VFEND®) — I.V charge dose 6 mg/kg/12h (2 doses) Maintenance iv treatment 4 mg/kg/12h during 6 days, followed by oral treatment (200 mg/12h)

SUMMARY:
Primary purpose: Frequency of use of broad-spectrum antifungals in the episode of neutropenia.

Secondary purposes:To determine the safety and toxicity measure by:

1. Frequency of Invader Fungal Infection.
2. Frequency of global use of broad-spectrum antifungals as amphotericine, itraconazole, voriconazole, caspofungin, terbinafine, during the period of study.
3. Mortality
4. Development of nephrotoxicity
5. Use of galactomannan in this clinical context
6. Time of administration of empirical antifungal therapy of broad-spectrum.

DETAILED DESCRIPTION:
Clinical trial with a pharmaceutical speciality in the conditions of authorized use

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients (from 2 years old on) with diagnostic of hematologic malignancies or solid tumour.
* Patients who will develop neutropenia (<500PN) post chemotherapy or post Bone Marrow Transplantation (BMT) that according to the center, they can receive empirical antifungal treatment of broad-spectrum.
* Controlled patients with galactomannan in blood twice weekly.
* Empirical antibacterial therapy of broad-spectrum, as possible the Pethema protocol that it is activated in this moment. Also it will be validated the monotherapy with carbapenemic or cephalosporin of fourth or third generation, or the biotherapy.
* Inclusion of patient since the start of his chemotherapy or therapy of preparation.
* If a bacterial infection is documented, it will be treated and controlled before to begin the empirical antifungal treatment.
* Signed of informed consent.
* Negative pregnancy test in fertile patients

Exclusion Criteria:

* Use of antifungal prophylaxis with triazoles with activity against Aspergillus, or use of others systematics antifungal by previous Invader Fungal Infection or other reasons.
* Use prophylactic of fluconazole to dose higher than 100 mg/day.
* Allergy to azoles
* To have a invader fungal infection at start of episode of neutropenia with fever.
* High effect in the unity of insulation of Candida strong to fluconazole that to opinion of center it hasn´t appropriate to include in a protocol where it is considered the use of empirical fluconazole.
* Neutropenias made by aplastic anemia or other faults of bone similar.
* Inclusion previous in this study.
* The patients will be excluded if they have settled by Aspergillus, C.krusei or C.gladiata in this episode of neutropenia, or in other and if they lack of the results of the cultures of vigilance in the present episode. If it presents positive result for any of those pathogens the empirical treatment will must be with a antifungal that it covers good (amphotericin, caspofungin or voriconazole) and not with fluconazole, then those patients will not follow this protocol.
* To receive drugs, which aren´t indicated in patients in treatment with voriconazole and/or with fluconazole.
* The patients will not be excluded if they receive antibacterial prophylaxis oral with quinolones, macrolides, etc., or stimulating factors G-CSF, GM-CSF or similar.
* Cause of exclusion will be the fault of fulfilment of inclusion criteria. Above all the patients will be excluded if they:
* have fault of twice weekly monitoring with galactomannan.
* have a bacterial infection not very good treated and controlled before to can begin the empirical antifungal infection (according to definition previous)
* have at final, a neutropenia of short stay that it has a risk important of Invader Fungal Infection. This data naturally will not know in the moment of include at patient in the study. It defines as neutropenia of short stay if it last out less of 5 days.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of use of broad-spectrum antifungals in the episode of neutropenia. | 2 years

SECONDARY OUTCOMES:
To determine the safety and toxicity measure by: | 1 year
Frequency of Invader Fungal Infection. | 2 years
Frequency of global use of broad-spectrum antifungals as amphotericine, itraconazole, voriconazole, caspofungin, terbinafine, during the period of study. | 2 years
Mortality | 2 years
Development of nephrotoxicity | 2 years
Use of galactomannan in this clinical context | 2 years
Time of administration of empirical antifungal therapy of broad-spectrum. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: de la Cámara Rafael, Dr, Principal Investigator — Hospital Universitario de la Princesa, Madrid
Locations (13):
- Spain (13):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Madrid
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Universitario Morales Meseguer, Murcia, Murcia, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Clínico Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Kami M, Machida U, Okuzumi K, Matsumura T, Mori Si S, Hori A, Kashima T, Kanda Y, Takaue Y, Sakamaki H, Hirai H, Yoneyama A, Mutou Y. Effect of fluconazole prophylaxis on fungal blood cultures: an autopsy-based study involving 720 patients with haematological malignancy. Br J Haematol. 2002 Apr;117(1):40-6. doi: 10.1046/j.1365-2141.2002.03414.x. PMID 11918531
- [Background] Young RC, Bennett JE, Vogel CL, Carbone PP, DeVita VT. Aspergillosis. The spectrum of the disease in 98 patients. Medicine (Baltimore). 1970 Mar;49(2):147-73. doi: 10.1097/00005792-197003000-00002. No abstract available. PMID 4913991
- [Background] Groll AH, Shah PM, Mentzel C, Schneider M, Just-Nuebling G, Huebner K. Trends in the postmortem epidemiology of invasive fungal infections at a university hospital. J Infect. 1996 Jul;33(1):23-32. doi: 10.1016/s0163-4453(96)92700-0. PMID 8842991
- [Background] Pizzo PA, Robichaud KJ, Gill FA, Witebsky FG. Empiric antibiotic and antifungal therapy for cancer patients with prolonged fever and granulocytopenia. Am J Med. 1982 Jan;72(1):101-11. doi: 10.1016/0002-9343(82)90594-0. No abstract available. PMID 7058815
- [Background] Empiric antifungal therapy in febrile granulocytopenic patients. EORTC International Antimicrobial Therapy Cooperative Group. Am J Med. 1989 Jun;86(6 Pt 1):668-72. doi: 10.1016/0002-9343(89)90441-5. PMID 2658574
- [Background] Wingard JR, Kubilis P, Lee L, Yee G, White M, Walshe L, Bowden R, Anaissie E, Hiemenz J, Lister J. Clinical significance of nephrotoxicity in patients treated with amphotericin B for suspected or proven aspergillosis. Clin Infect Dis. 1999 Dec;29(6):1402-7. doi: 10.1086/313498. PMID 10585786
- [Background] Bates DW, Su L, Yu DT, Chertow GM, Seger DL, Gomes DR, Dasbach EJ, Platt R. Mortality and costs of acute renal failure associated with amphotericin B therapy. Clin Infect Dis. 2001 Mar 1;32(5):686-93. doi: 10.1086/319211. Epub 2001 Feb 21. PMID 11229835
- [Background] Harbarth S, Burke JP, Lloyd JF, Evans RS, Pestotnik SL, Samore MH. Clinical and economic outcomes of conventional amphotericin B-associated nephrotoxicity. Clin Infect Dis. 2002 Dec 15;35(12):e120-7. doi: 10.1086/344468. Epub 2002 Dec 2. PMID 12471588
- [Background] Walsh TJ, Teppler H, Donowitz GR, Maertens JA, Baden LR, Dmoszynska A, Cornely OA, Bourque MR, Lupinacci RJ, Sable CA, dePauw BE. Caspofungin versus liposomal amphotericin B for empirical antifungal therapy in patients with persistent fever and neutropenia. N Engl J Med. 2004 Sep 30;351(14):1391-402. doi: 10.1056/NEJMoa040446. PMID 15459300
- [Background] Walsh TJ, Pappas P, Winston DJ, Lazarus HM, Petersen F, Raffalli J, Yanovich S, Stiff P, Greenberg R, Donowitz G, Schuster M, Reboli A, Wingard J, Arndt C, Reinhardt J, Hadley S, Finberg R, Laverdiere M, Perfect J, Garber G, Fioritoni G, Anaissie E, Lee J; National Institute of Allergy and Infectious Diseases Mycoses Study Group. Voriconazole compared with liposomal amphotericin B for empirical antifungal therapy in patients with neutropenia and persistent fever. N Engl J Med. 2002 Jan 24;346(4):225-34. doi: 10.1056/NEJM200201243460403. PMID 11807146
- [Background] Malik IA, Moid I, Aziz Z, Khan S, Suleman M. A randomized comparison of fluconazole with amphotericin B as empiric anti-fungal agents in cancer patients with prolonged fever and neutropenia. Am J Med. 1998 Dec;105(6):478-83. doi: 10.1016/s0002-9343(98)00326-x. PMID 9870832
- [Background] Viscoli C, Castagnola E, Van Lint MT, Moroni C, Garaventa A, Rossi MR, Fanci R, Menichetti F, Caselli D, Giacchino M, Congiu M. Fluconazole versus amphotericin B as empirical antifungal therapy of unexplained fever in granulocytopenic cancer patients: a pragmatic, multicentre, prospective and randomised clinical trial. Eur J Cancer. 1996 May;32A(5):814-20. doi: 10.1016/0959-8049(95)00619-2. PMID 9081359
- [Background] Winston DJ, Hathorn JW, Schuster MG, Schiller GJ, Territo MC. A multicenter, randomized trial of fluconazole versus amphotericin B for empiric antifungal therapy of febrile neutropenic patients with cancer. Am J Med. 2000 Mar;108(4):282-9. doi: 10.1016/s0002-9343(99)00457-x. PMID 11014720
- [Background] McLintock LA, Jordanides NE, Allan EK, Copland M, Stewart K, Parker A, Devaney M, Holyoake TL, Jones BL. The use of a risk group stratification in the management of invasive fungal infection: a prospective validation. Br J Haematol. 2004 Feb;124(3):403-4. doi: 10.1046/j.1365-2141.2003.04794.x. No abstract available. PMID 14717790
- [Background] Wheat LJ. Rapid diagnosis of invasive aspergillosis by antigen detection. Transpl Infect Dis. 2003 Dec;5(4):158-66. doi: 10.1111/j.1399-3062.2003.00031.x. PMID 14987199
- [Background] Mennink-Kersten MA, Donnelly JP, Verweij PE. Detection of circulating galactomannan for the diagnosis and management of invasive aspergillosis. Lancet Infect Dis. 2004 Jun;4(6):349-57. doi: 10.1016/S1473-3099(04)01045-X. PMID 15172343
- [Background] Herbrecht R, Letscher-Bru V, Oprea C, Lioure B, Waller J, Campos F, Villard O, Liu KL, Natarajan-Ame S, Lutz P, Dufour P, Bergerat JP, Candolfi E. Aspergillus galactomannan detection in the diagnosis of invasive aspergillosis in cancer patients. J Clin Oncol. 2002 Apr 1;20(7):1898-906. doi: 10.1200/JCO.2002.07.004. PMID 11919250
- [Background] Maertens J, Theunissen K, Verbeken E, Lagrou K, Verhaegen J, Boogaerts M, Eldere JV. Prospective clinical evaluation of lower cut-offs for galactomannan detection in adult neutropenic cancer patients and haematological stem cell transplant recipients. Br J Haematol. 2004 Sep;126(6):852-60. doi: 10.1111/j.1365-2141.2004.05140.x. PMID 15352990
- [Background] Marr KA, Balajee SA, McLaughlin L, Tabouret M, Bentsen C, Walsh TJ. Detection of galactomannan antigenemia by enzyme immunoassay for the diagnosis of invasive aspergillosis: variables that affect performance. J Infect Dis. 2004 Aug 1;190(3):641-9. doi: 10.1086/422009. Epub 2004 Jul 1. PMID 15243943
- [Background] Viscoli C, Machetti M, Cappellano P, Bucci B, Bruzzi P, Van Lint MT, Bacigalupo A. False-positive galactomannan platelia Aspergillus test results for patients receiving piperacillin-tazobactam. Clin Infect Dis. 2004 Mar 15;38(6):913-6. doi: 10.1086/382224. Epub 2004 Feb 27. PMID 14999640
- [Background] Singh N, Obman A, Husain S, Aspinall S, Mietzner S, Stout JE. Reactivity of platelia Aspergillus galactomannan antigen with piperacillin-tazobactam: clinical implications based on achievable concentrations in serum. Antimicrob Agents Chemother. 2004 Jun;48(6):1989-92. doi: 10.1128/AAC.48.6.1989-1992.2004. PMID 15155189
- [Background] Sulahian A, Boutboul F, Ribaud P, Leblanc T, Lacroix C, Derouin F. Value of antigen detection using an enzyme immunoassay in the diagnosis and prediction of invasive aspergillosis in two adult and pediatric hematology units during a 4-year prospective study. Cancer. 2001 Jan 15;91(2):311-8. doi: 10.1002/1097-0142(20010115)91:23.0.co;2-3. PMID 11180076
- [Background] Maertens J, Van Eldere J, Verhaegen J, Verbeken E, Verschakelen J, Boogaerts M. Use of circulating galactomannan screening for early diagnosis of invasive aspergillosis in allogeneic stem cell transplant recipients. J Infect Dis. 2002 Nov 1;186(9):1297-306. doi: 10.1086/343804. Epub 2002 Oct 8. PMID 12402199
- [Background] Heussel CP, Kauczor HU, Heussel GE, Fischer B, Begrich M, Mildenberger P, Thelen M. Pneumonia in febrile neutropenic patients and in bone marrow and blood stem-cell transplant recipients: use of high-resolution computed tomography. J Clin Oncol. 1999 Mar;17(3):796-805. doi: 10.1200/JCO.1999.17.3.796. PMID 10071269
- [Background] Ascioglu S, Rex JH, de Pauw B, Bennett JE, Bille J, Crokaert F, Denning DW, Donnelly JP, Edwards JE, Erjavec Z, Fiere D, Lortholary O, Maertens J, Meis JF, Patterson TF, Ritter J, Selleslag D, Shah PM, Stevens DA, Walsh TJ; Invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Mycoses Study Group of the National Institute of Allergy and Infectious Diseases. Defining opportunistic invasive fungal infections in immunocompromised patients with cancer and hematopoietic stem cell transplants: an international consensus. Clin Infect Dis. 2002 Jan 1;34(1):7-14. doi: 10.1086/323335. Epub 2001 Nov 26. PMID 11731939
- [Background] Walsh TJ, Finberg RW, Arndt C, Hiemenz J, Schwartz C, Bodensteiner D, Pappas P, Seibel N, Greenberg RN, Dummer S, Schuster M, Holcenberg JS. Liposomal amphotericin B for empirical therapy in patients with persistent fever and neutropenia. National Institute of Allergy and Infectious Diseases Mycoses Study Group. N Engl J Med. 1999 Mar 11;340(10):764-71. doi: 10.1056/NEJM199903113401004. PMID 10072411
- [Background] Sociedad Espanola de Quimioterapia; Asociacion Espanola de Hematologia y Hemoterapia. [Prophylaxis and treatment of fungal infections in oncohematological patients]. Rev Esp Quimioter. 2002 Dec;15(4):387-401. No abstract available. Spanish. PMID 12607556
- [Background] Herbrecht R, Denning DW, Patterson TF, Bennett JE, Greene RE, Oestmann JW, Kern WV, Marr KA, Ribaud P, Lortholary O, Sylvester R, Rubin RH, Wingard JR, Stark P, Durand C, Caillot D, Thiel E, Chandrasekar PH, Hodges MR, Schlamm HT, Troke PF, de Pauw B; Invasive Fungal Infections Group of the European Organisation for Research and Treatment of Cancer and the Global Aspergillus Study Group. Voriconazole versus amphotericin B for primary therapy of invasive aspergillosis. N Engl J Med. 2002 Aug 8;347(6):408-15. doi: 10.1056/NEJMoa020191. PMID 12167683
- [Background] Pfaller MA, Diekema DJ; International Fungal Surveillance Participant Group. Twelve years of fluconazole in clinical practice: global trends in species distribution and fluconazole susceptibility of bloodstream isolates of Candida. Clin Microbiol Infect. 2004 Mar;10 Suppl 1:11-23. doi: 10.1111/j.1470-9465.2004.t01-1-00844.x. PMID 14748799
- [Background] Pappas PG, Rex JH, Sobel JD, Filler SG, Dismukes WE, Walsh TJ, Edwards JE; Infectious Diseases Society of America. Guidelines for treatment of candidiasis. Clin Infect Dis. 2004 Jan 15;38(2):161-89. doi: 10.1086/380796. Epub 2003 Dec 19. No abstract available. PMID 14699449
- [Background] Goodman JL, Winston DJ, Greenfield RA, Chandrasekar PH, Fox B, Kaizer H, Shadduck RK, Shea TC, Stiff P, Friedman DJ, et al. A controlled trial of fluconazole to prevent fungal infections in patients undergoing bone marrow transplantation. N Engl J Med. 1992 Mar 26;326(13):845-51. doi: 10.1056/NEJM199203263261301. PMID 1542320
- [Background] Winston DJ, Chandrasekar PH, Lazarus HM, Goodman JL, Silber JL, Horowitz H, Shadduck RK, Rosenfeld CS, Ho WG, Islam MZ, Buell DN. Fluconazole prophylaxis of fungal infections in patients with acute leukemia. Results of a randomized placebo-controlled, double-blind, multicenter trial. Ann Intern Med. 1993 Apr 1;118(7):495-503. doi: 10.7326/0003-4819-118-7-199304010-00003. PMID 8442620
- [Background] Rotstein C, Bow EJ, Laverdiere M, Ioannou S, Carr D, Moghaddam N. Randomized placebo-controlled trial of fluconazole prophylaxis for neutropenic cancer patients: benefit based on purpose and intensity of cytotoxic therapy. The Canadian Fluconazole Prophylaxis Study Group. Clin Infect Dis. 1999 Feb;28(2):331-40. doi: 10.1086/515128. PMID 10064252
- [Background] Wolff SN, Fay J, Stevens D, Herzig RH, Pohlman B, Bolwell B, Lynch J, Ericson S, Freytes CO, LeMaistre F, Collins R, Pineiro L, Greer J, Stein R, Goodman SA, Dummer S. Fluconazole vs low-dose amphotericin B for the prevention of fungal infections in patients undergoing bone marrow transplantation: a study of the North American Marrow Transplant Group. Bone Marrow Transplant. 2000 Apr;25(8):853-9. doi: 10.1038/sj.bmt.1702233. PMID 10808206
- [Background] Slavin MA, Osborne B, Adams R, Levenstein MJ, Schoch HG, Feldman AR, Meyers JD, Bowden RA. Efficacy and safety of fluconazole prophylaxis for fungal infections after marrow transplantation--a prospective, randomized, double-blind study. J Infect Dis. 1995 Jun;171(6):1545-52. doi: 10.1093/infdis/171.6.1545. PMID 7769290
- [Background] MacMillan ML, Goodman JL, DeFor TE, Weisdorf DJ. Fluconazole to prevent yeast infections in bone marrow transplantation patients: a randomized trial of high versus reduced dose, and determination of the value of maintenance therapy. Am J Med. 2002 Apr 1;112(5):369-79. doi: 10.1016/s0002-9343(01)01127-5. PMID 11904111
- [Background] Marr KA, Crippa F, Leisenring W, Hoyle M, Boeckh M, Balajee SA, Nichols WG, Musher B, Corey L. Itraconazole versus fluconazole for prevention of fungal infections in patients receiving allogeneic stem cell transplants. Blood. 2004 Feb 15;103(4):1527-33. doi: 10.1182/blood-2003-08-2644. Epub 2003 Oct 2. PMID 14525770
- See also: Spanish association of Haematology — http://www.aehh.org